CLINICAL TRIAL: NCT01383863
Title: A Prospective Observational Study Cohort to Assess the Rate of Castration Resistance, Disease Progression and Overall Survival Over a 3-year Period Post-androgen Deprivation Therapy Induction in Patients With Advanced Prostate Cancer Who Have Previously Participated in the Triptocare Study (Http://Clinicaltrials.Gov/ct2/Show/Study/NCT01020448)
Brief Title: A Long-term Observational Study Cohort in Patients With Advanced Prostate Cancer
Acronym: TRIPTOCARE LT
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-52014-187
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to assess the rate of castration resistance, disease progression and overall survival over a 3-year period post-androgen deprivation therapy (ADT) induction in a study cohort of patients with advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Have participated and received study treatment in the Triptocare study
* Be aware of the investigational nature of this observational study cohort and must give written (personally signed and dated) informed consent

Exclusion Criteria:

* Absence of written informed consent from the patient

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously diagnosed advanced prostate cancer, and who have participated in the Triptocare study and who have given written informed consent to participate in the study. They have therefore been treated with triptorelin (22.5 mg, intamuscular) as an ADT induction.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Castration-resistant prostate cancer (CRPC) | Over a 3-year period post-androgen deprivation therapy induction

SECONDARY OUTCOMES:
Disease progression (DP) rate post-androgen deprivation therapy induction | Over a 3-year period post-androgen deprivation therapy induction
Overall survival | 3-years post-androgen deprivation therapy induction
Serum prostate specific antigen | Over a 3-year period post-androgen deprivation therapy induction
Serum testosterone | Over a 3-year period post-androgen deprivation therapy induction

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (35):
- Denmark (4):
  - Fredericia Sygehus, Fredericia
  - Frederiksbergs Hospital, Frederiksberg
  - Herlev University Hospital, Herlev
  - Odense Universitets Hospital, Odense
- France (13):
  - Clinique Rhône Durance, Avignon
  - Hôpital Pellegrin, Bordeaux
  - CHU Henri Mondor, Créteil
  - Chru Lille, Lille
  - Hôpital Nord, Marseille
  - Clinique Beau Soleil, Montpellier
  - Private practice, Nancy
  - CHU Nantes, Nantes
  - CHU Pasteur, Nice
  - Hôpital Val de Grâce, Paris
  - Institut Mutualiste Monsouris, Paris
  - Hôpital Henry Gabrielle, Saint-Genis-Laval
  - Hôpital Foch, Suresnes
- Latvia (2):
  - P.Stradins Clinical University Hospital, Riga
  - Center of Oncology, Riga
- Lithuania (3):
  - Medical University Clinics, Kaunas
  - University Hospital, Klaipėda
  - University Oncological Institute, Vilnius
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Diaconessenhuis, Leiden
- Romania (3):
  - Medical Center, Arad
  - Sc E-Uro Srl, Cluj-Napoca
  - Oncomed, Timișoara
- United Kingdom (8):
  - Ulster hospital, Belfast
  - Bristol Royal Infirmary, Bristol
  - Addenbrookes Hospital, Cambridge
  - University Hospital Wales, Cardiff
  - University Hospital Coventry, Coventry
  - Leicester General Hospital, Leicester
  - Nottingham City Hospital, Nottingham
  - Lister Hospital, Stevenage

REFERENCES:
- See also: Triptocare study NCT01020448 — http://clinicaltrials.gov/ct2/show/study/NCT01020448